CLINICAL TRIAL: NCT00997308
Title: A Phase I, Randomised, Double-blind, Placebo-controlled, Parallel Group, Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD1446 in Healthy Elderly Male and Female Volunteers During 4 Weeks of Treatment
Brief Title: A Study to Investigate Safety, Tolerability and Pharmacokinetics of AZD1446 Administered for 4 Weeks in Elderly Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D1950C00009; EudraCT No.2009-013390-18
Record Dates: First submitted 2009-10-12; First posted 2009-10-19 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: AZD1446; to investigate safety and tolerability in Healthy subjects during 4 weeks of administration
MeSH Terms: interventions — 3-(5-chloro-2-furoyl)-3,7-diazabicyclo(3.3.0)octane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD1446 Low (Experimental): Low dose of AZD1446
  Interventions: Drug: AZD1446
- AZD1446 High (Experimental): High dose of AZD1446
  Interventions: Drug: AZD1446
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1446 — Solution, oral, for 4 weeks
  Arms: AZD1446 High; AZD1446 Low
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety, tolerability and pharmacokinetics (PK) of two doses of AZD1446 or placebo in subjects when given for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-fertile female, elderly Subjects, aged ≥65 to ≤85
* Body mass index (BMI) between 18 and 30 kg/m2
* Clinically normal findings on physical examination

Exclusion Criteria:

* History of any clinically significant disease or disorder
* History of severe allergy/hypersensitivity reactions including severe food allergy as judged by the investigator.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 97 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of AZD1446 dosed for 4 weeks as compared to placebo in healthy elderly male and female volunteers. Safety and tolerability outcomes include adverse events, clinical chemistry and vitals (pulse and blood pressure). | During the whole study period, Study days 1-68 (30 days of enrolment , study day 1-28 and follow up visit study days 35-38).

SECONDARY OUTCOMES:
To determine the PK of AZD1446 dosed for 4 weeks in healthy elderly male and female volunteers. PK parameters include renal clearance, AUC (0-24)ss and T1/2 eff. | PK sampling taken at defined timepoints during the treatment period (study days 1-28)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Fransson, MD, PhD, Principal Investigator — AstraZeneca R&DClinical Pharmacology Unit CPUTunavägen 22aS-221 87 LundSweden; Björn Paulsson, MD, PhD, Study Director — AstraZeneca R&D SödertäljeSE-151 85 SödertäljeSweden
Locations (1):
- Research, Lund, Sweden